CLINICAL TRIAL: NCT06449560
Title: Department of Physical Medicine and Rehabilitation, Wang Fang Hospital, Taipei Medical University, Taipei, Taiwan
Brief Title: Applying Videos Feedback Learning to Improve Skills Performance of Physiotherapy Interns
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, I Hsien Lin, Clinical Professor, Taipei Medical University WanFang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: N202211059
Record Dates: First submitted 2023-12-10; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Feedback
Keywords: Videos Feedback; Skills Performance; Physiotherapy
MeSH Terms: interventions — Group Practice

STUDY DESIGN:
Intervention Model Description: Randomized, single-blinded, two parallel-groups trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Practice Group (Active Comparator): Participants in this group engage in the traditional core course, followed by a 20-minute practical session where they pair up for mutual hands-on practice. The assessment of upper limb soft tissue operations takes approximately 4 minutes per session, allowing for approximately 5 practice sessions.
  Interventions: Other: Practice Group
- Video Feedback Group (Experimental): Participants receive the traditional core course along with a 20-minute video feedback session. Initially, a therapist records students' assessment techniques in action, capturing the dynamic process on video. The recorded video is then played on a screen for both the course teacher and students to watch together. Participants can annotate specific actions during the viewing, and the course teacher facilitates a reflective discussion where participants observe and identify any issues or correct actions as expected. The teacher provides feedback on areas of improvement in the action process for further practice. The self-viewing of the recorded video serves as a valuable tool for enhancing the skill performance of physical therapy interns.
  Interventions: Other: Practice Group; Other: Video Feedback Group

INTERVENTIONS:
Other: Practice Group — Participants in this group engage in the traditional core course (1-hour lecture on upper limb soft tissue differential diagnosis and assessment techniques. They have the opportunity to observe teacher demonstrations, and the course content and instructional demonstrations are consistent and delivered by the same therapist), followed by a 20-minute practical session where they pair up for mutual hands-on practice. The assessment of upper limb soft tissue operations takes approximately 4 minutes per session, allowing for approximately 5 practice sessions.
Other: Video Feedback Group — Participants receive the traditional core course (as the same in the practice group) along with a 20-minute video feedback session. Initially, a therapist records students' assessment techniques in action, capturing the dynamic process on video. The recorded video is then played on a screen for both the course teacher and students to watch together. Participants can annotate specific actions during the viewing, and the course teacher facilitates a reflective discussion where participants observe and identify any issues or correct actions as expected. The teacher provides feedback on areas of improvement in the action process for further practice. The self-viewing of the recorded video serves as a valuable tool for enhancing the skill performance of physical therapy interns.
  Arms: Video Feedback Group

SUMMARY:
This project uses self-practicing videos feedback to learn to improve the skill performance of physiotherapy interns. For traditional physiotherapy intern courses, teachers will conduct core courses and demonstrate teaching, but students are less familiar with the application of skills, even if adding practice course. The learning outcomes of the course are still not good in skill performance. By recording the self-practicing videos, the teacher uses observation and feedback to let the physiotherapy interns know whether the posture of the individual case, the fixed position of the limbs are appropriate, the resistance given and whether the verbal instruction is correct, and based on the evaluation outcomes to observe the students' learning status and clinical thinking ability can improve the skill performance and learning satisfaction.

DETAILED DESCRIPTION:
Methods:

A parallel-group design. Ninety physiotherapy interns from a medical institution were enrolled as participants, with practice and videos feedback groups each comprising 45 participants. Two groups received traditional core course. The practice group received an additional 20 minutes of practice course. However, the videos feedback group received an additional 20 minutes of recording the self-practicing videos, the teacher uses observation and feedback learning of evaluation skills to improve the performance of physical therapy interns.The Direct Observation of Procedural Skills, Mini-Clinical Evaluation Exercise, Objective structured clinical examination, and satisfaction questionnaire were used in a pretest, posttest and the follow-up test.The inclusion criteria was being older than 20 years.Students were excluded if they could not complete the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* physical therapy interns require individuals to be over 20 years old.

Exclusion Criteria:

* Individuals unwilling to participate in the study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Objective Structured Clinical Examination (OSCE) | pre-test, within 1 week post test, 3-month follow-up
  Evaluators utilize a detailed, operationally defined standardized checklist to assess the performance of examinees in a structured clinical skills assessment. This instructional design aims to aid students in learning and understanding their learning outcomes, evaluating the knowledge, skills, and attitudes of the examinees through a performance-based testing approach.
  The scoring sheet includes an standardized checklist and an overall performance assessment. The standardized checklist comprises 15 items, with results presented in percentages, where higher scores indicate better performance. The overall performance assessment ranges from 5 points (excellent) to 1 point (poor).

SECONDARY OUTCOMES:
Mini-Clinical Evaluation Exercise (Mini-CEX) | pre-test, within 1 week post test, 3-month follow-up
  The Mini-CEX focuses on the performance of interactions with patients. Clinical instructors can use it to directly observe the interaction between learners and patients, conduct a simple assessment of the Mini-CEX, and provide direct feedback to the learners. Clinical instructors can assess a specific aspect (medical interview, physical examination, operational skills, counseling and health education, clinical judgment, organizational efficiency, humanitarian professionalism) each time.
  The assessment consists of 7 items, with scores ranging from 1 to 9 points each. The total score ranges from 7 to 63 points, with higher scores indicating better performance.
Direct Observation of Procedural Skills (DOPS) | pre-test, within 1 week post test, 3-month follow-up
  Clinical instructors evaluate and provide feedback on the procedural skills of the examinee. Each clinical procedural skill is assessed and feedback is provided to ensure learning effectiveness.
  The assessment consists of 10 items, with scores ranging from 1 to 6 points each. The total score ranges from 10 to 60 points, with higher scores indicating better performance.
Course Satisfaction | within 1 week post test
  Understand your satisfaction with various arrangements of this course activity, including speakers, lecture content, and related activities.
  The assessment consists of 12 items, with scores ranging from 1 to 5 points each. The total score ranges from 12 to 60 points, with higher scores indicating higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Hsien I Lin, MS, Principal Investigator — Wan Fang Hospital, Taipei Medical University

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol, Statistical Analysis Plan, Clinical Study Report
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Individual Participant Data Sharing Plan Description Data will last for 3 years after the end of the study.
Access Criteria: Ecxel

REFERENCES:
- [Background] Miller GE. The assessment of clinical skills/competence/performance. Acad Med. 1990 Sep;65(9 Suppl):S63-7. doi: 10.1097/00001888-199009000-00045. No abstract available. PMID 2400509
- [Background] Mori B, Carnahan H, Herold J. Use of Simulation Learning Experiences in Physical Therapy Entry-to-Practice Curricula: A Systematic Review. Physiother Can. 2015 Spring;67(2):194-202. doi: 10.3138/ptc.2014-40E. PMID 25931672
- [Background] Blackstock FC, Watson KM, Morris NR, Jones A, Wright A, McMeeken JM, Rivett DA, O'Connor V, Peterson RF, Haines TP, Watson G, Jull GA. Simulation can contribute a part of cardiorespiratory physiotherapy clinical education: two randomized trials. Simul Healthc. 2013 Feb;8(1):32-42. doi: 10.1097/SIH.0b013e318273101a. PMID 23250189
- [Background] Watson K, Wright A, Morris N, McMeeken J, Rivett D, Blackstock F, Jones A, Haines T, O'Connor V, Watson G, Peterson R, Jull G. Can simulation replace part of clinical time? Two parallel randomised controlled trials. Med Educ. 2012 Jul;46(7):657-67. doi: 10.1111/j.1365-2923.2012.04295.x. Epub 2012 May 30. PMID 22646319
- [Background] Sanders BR, Ruvolo JF. Mock clinic. An approach to clinical education. Phys Ther. 1981 Aug;61(8):1163-7. doi: 10.1093/ptj/61.8.1163. PMID 7267707
- [Background] Guadagnoli MA, Lee TD. Challenge point: a framework for conceptualizing the effects of various practice conditions in motor learning. J Mot Behav. 2004 Jun;36(2):212-24. doi: 10.3200/JMBR.36.2.212-224. PMID 15130871
- [Background] Emmen HH, Wesseling LG, Bootsma RJ, Whiting HT, Van Wieringen PC. The effect of video-modelling and video-feedback on the learning of the tennis service by novices. J Sports Sci. 1985 Summer;3(2):127-38. doi: 10.1080/02640418508729742. PMID 4094023
- [Background] Wulf G, Shea C, Lewthwaite R. Motor skill learning and performance: a review of influential factors. Med Educ. 2010 Jan;44(1):75-84. doi: 10.1111/j.1365-2923.2009.03421.x. PMID 20078758
- [Background] Duffy A. A concept analysis of reflective practice: determining its value to nurses. Br J Nurs. 2007 Dec 13-2008 Jan 9;16(22):1400-7. doi: 10.12968/bjon.2007.16.22.27771. PMID 18361389
- [Background] Rotthoff T, Ostapczuk MS, Kroncke KD, Zimmerhofer A, Decking U, Schneider M, Ritz-Timme S. Criterion validity of a competency-based assessment center in medical education--a 4-year follow-up study. Med Educ Online. 2014 Sep 12;19:25254. doi: 10.3402/meo.v19.25254. eCollection 2014. PMID 25219931

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-04): https://cdn.clinicaltrials.gov/large-docs/60/NCT06449560/Prot_SAP_000.pdf